CLINICAL TRIAL: NCT06967909
Title: Effectiveness of Tai Chi and Acupuncture in the Prophylaxes of Episodic Migraine in Hong Kong Chinese Women and the Analysis of Microstructural White Matter Alterations: a Non-inferiority Single-blind Randomized Controlled Trial
Brief Title: Effectiveness of Tai Chi and Acupuncture on Migraine Attack Prevention and Brain White Matter Changes: A Non-Inferiority RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23B2-029A
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Migraine; Migraine Disorder
Keywords: Migraine; Tai Chi; Acupuncture; Women; Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi training (Experimental): Participants in this arm will receive 24-week Tai Chi training. F
  Interventions: Behavioral: Tai Chi training
- Acupuncture (Active Comparator): Participants in this arm will receive 30 sessions of acupuncture treatment over a period of 24 weeks.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Behavioral: Tai Chi training — Participants will receive 24 weeks of Tai Chi training. For the first 12 weeks, they will receive 3 instructor-led Tai Chi training sessions per week, and practice 2 Tai Chi sessions by themselves. In the next 12 weeks, they will receive 1 instructor-led Tai Chi session and self-practice 2 Tai Chi sessions per week. A modified 33-short form Yang-style Tai Chi Chuan will be adopted. The Tai Chi sessions will be operated by qualified instructors. Each 1-hour training session consists of 10 minutes brief warm-up stretching session followed by 45 minutes standard Tai Chi routine activities, and 5 minutes of cool-down stretching. The Tai Chi instructors are required to attend a training session that ensure all of them to deliver the same intervention protocol throughout the study. The research assistant will monitor the fidelity of intervention by visiting the Tai Chi sessions frequently. The training session will be delivered in group. The group size is 25-30 persons.
  Arms: Tai Chi training
Procedure: Acupuncture — Participants in the acupuncture group will receive 30 acupuncture treatment sessions, each last for 1 hour. Acupuncture will be performed every 2 days within one week, followed by a 3-day break, i.e., twice a week for the first 12 weeks; then it will be performed once every two weeks for the next 12 weeks. In total 30 sessions during 24 weeks treatment period. All acupuncture sessions will be administered by registered Traditional Chinese Medicine practitioners in Hong Kong with at least three years of clinical experience.
  Arms: Acupuncture

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of Tai Chi training and acupuncture on the migraine attacks and structural brain changes in women with episodic migraine.

Researchers will compare Tai Chi training to acupuncture treatment in a randomized controlled trial with 132 female participants. Participants will:

* Be randomly assigned to either the Tai Chi group or the acupuncture group.
* Undergo a 24-week intervention, with structured sessions for Tai Chi or scheduled acupuncture treatments.
* Complete assessments through migraine diaries, questionnaires, physical measurements, MRI and TCD scans at various time points.

The study ensures participant safety through close monitoring, with medical support available in case of discomfort. Data confidentiality will be maintained, with encrypted storage and restricted access for research purposes.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine whether Tai Chi training has the similar effectiveness in reducing the frequency of migraine attacks as acupuncture; and whether both Tai Chi and acupuncture can improve structural brain changes in women with episodic migraine. It also aims to examine whether the improvements in migraine features are linked to the structural brain changes and better cerebrovascular function after the intervention.

This study is a randomized controlled trial with 132 women who have episodic migraines. Participants will be randomly assigned to either the Tai Chi training group or the acupuncture treatment group, with 66 individuals in each group.

Participants will:

* receive a 24-week intervention, which the Tai Chi group attends instructor-led training sessions and self-practice sessions, and the acupuncture group receives 30 treatment sessions over the same period.
* Undergo assessments, including migraine diaries for migraine features and symptoms; migraine characteristics, lifestyle factors, body measurements (e.g., height, weight, and body composition), and advanced imaging techniques including MRI and TCD scans.
* Data will be collected at baseline, the 12th week, and the 24th week. MRI will be used to assess white matter changes, while TCD will be used to evaluate cerebrovascular function. Both procedures are safe and non-invasive, with specific pre-exam precautions.

To ensure participant safety, Tai Chi sessions will be closely monitored for any adverse effects such as dizziness or falls, while acupuncture treatments will be supervised to address any discomfort. If participants experience intolerable migraines, they will receive guided medication management.

Confidentiality will be strictly maintained, with encrypted data storage and restricted access for research auditing. Personal identifiers will not be linked to the data, and all records will be securely stored for five years before being destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women aged 18 years and above;
* Diagnosed with episodic migraines, with or without aura, according to the International Classification of Headache Disorders, 3rd edition (ICHD-3);
* Migraine attack frequency ranging from 2 to 14 days per month (≥15 days/month is classified as chronic migraine and is not included in this study);
* Assessed by a sports specialist as capable of engaging in moderate physical activity;
* Residing in Hong Kong.

Exclusion Criteria:

* Unable to engage in moderate physical activity;
* Comorbid with other neurological disorders;
* Experiencing non-migraine headaches for more than 5 days per month;
* Previous practice of Tai Chi or other mind-body exercises (such as yoga, biofeedback, meditation, etc.);
* Received alternative treatments for migraines (such as acupuncture or Chinese medicine) during the recruitment period or within the past 12 weeks;
* Undergoing preventive medication treatment for migraines during the recruitment period or within the past 12 weeks;
* Excessive use of medication, taking antipsychotic or antidepressant drugs, or using analgesics for other chronic pain conditions for more than 3 days per month within the past 12 weeks;
* Diagnosed with epilepsy or having a mental illness;
* Pregnant, breastfeeding, or currently taking contraceptive medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The difference in frequency of migraine attacks | Between 4 weeks before randomization and weeks 9-12 / 21-24 after randomization
  The frequency of migraine attacks will be measured by the number of attacks per month.
The difference in migraine days | Between 4 weeks before randomization and weeks 9-12 / 21-24 after randomization
  The frequency of migraine days will be measured by the days with migraine attacks per month.
The difference of white matter abnormalities (WMAs) | From the baseline to 24 weeks
  All the participants in the Tai Chi group will be measured with MRI. The appearance, number, size and location of WMAs will be recorded. Two experienced neurologists or neuroradiologists will be invited to review the MRI scans independently. Scheltens' visual rating scale will be used to measure the degree of WMAs. Briefly, WMAs will be separately graded in each of the following locations: frontal lobes, temporal lobes, parietal lobes and occipital lobes. WMAs will be graded as follows: 0 (no lesions), 1 (hyperintensity < 3 mm and n ≤ 5), 2 (< 3 mm and n ≥ 6), 3 (4-10 mm and n ≤ 5), 4 (4-10 mm and n ≥ 6), 5 (≥ 11 mm and n ≥ 1), and 6 (confluent). The sum of scores from each location will be considered as the final score. Only the women who are identified WMAs (Scheltens' visual rating scores >0) will take the MRI test again at the 24th week.

SECONDARY OUTCOMES:
The proportion of responders | From the baseline to 12 weeks and 24 weeks
  Defined as the proportion of patients with at least a 50% reduction of the number of attacks per month.
The intensity of the headache | From the baseline to 12 weeks and 24 weeks
  The intensity of the headache measured by a Visual Analogue Scale (VAS). This scale is most commonly anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10). Higher scores indicate higher level of headache intensity.
The duration of headache | From the baseline to 12 weeks and 24 weeks
  The duration of headache recorded in the migraine diary to the nearest 0.1 hour.
Migraine related disability | From the baseline to 12 weeks and 24 weeks
  Migraine related disability measured by the Migraine Disability Assessment Score (MIDAS). The MIDAS consists of five items that reflect the number of days reported as either missing or with reduced productivity at work, home, and social events in last 3 months and two additional items that assess the number of days with headaches in the last 3 months and a scale of the painfulness of the headaches. The MIDAS is scored as the sum of days reported in the first five questions. Higher scores are indicative of more disability.
Stress level | From the baseline to 12 weeks and 24 weeks
  Stress level evaluated by the Perceived Stress Scale-14 (PSS-14). The total score of PSS-14 ranges from 0 to 56 with higher scores indicating higher perceived stress.
Sleep quality | From the baseline to 12 weeks and 24 weeks
  Sleep quality examined by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). The global score of PSQI ranges from 0 to 21 with a higher score indicating worse sleep quality.
Fatigue level | From the baseline to 12 weeks and 24 weeks
  Fatigue level evaluated by the Numeric Rating Scale-fatigue scale (NRS). NRS evaluates fatigue level at a 0-to-10 scale, with 0 indicating no fatigue and 10 indicating the worst possible fatigue.
Health related Quality-of-Life | From the baseline to 12 weeks and 24 weeks
  Health related Quality-of-Life measured by the Migraine-Specific Quality-of-Life Questionnaire (MSQ). The total scores of MSQ range from 0-100, with a higher score indicating better Quality-of-Life.
Weight | From the baseline to 12 weeks and 24 weeks
  Weight in kilograms
Height | From the baseline to 12 weeks and 24 weeks
  Height in meters
Waist circumference | From the baseline to 12 weeks and 24 weeks
  Waist circumference in centimeter
Hip circumference | From the baseline to 12 weeks and 24 weeks
  Hip circumference in centimeter
Percent body fat | From the baseline to 12 weeks and 24 weeks
  Percent body fat in %
The difference of pulsatility index (PI) | From the baseline to 12 weeks and 24 weeks
  PI in neck vessels will be measured and recorded by Transcranial Doppler (TCD).
The difference of mean blood flow velocity (MBFV) | From the baseline to 12 weeks and 24 weeks
  MBFV in neck vessels will be measured and recorded by Transcranial Doppler (TCD).
The difference of impaired cerebrovascular responsiveness (CVR) | From the baseline to 12 weeks and 24 weeks
  CVR in neck vessels will be measured and recorded by Transcranial Doppler (TCD).

CONTACTS AND LOCATIONS:
Overall Officials: Yao Jie Xie, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No